CLINICAL TRIAL: NCT00087035
Title: Phase II Trial Of TAXOTERE + TARCEVA™ To Treat HRPC In Men ≥ 65 Years Of Age
Brief Title: Docetaxel and Erlotinib in Treating Older Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Genentec (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000372833; UCLA-0308082; AVENTIS-GIA-16115; GENENTECH-OSI-2527S
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Taxotere plus Tarceva (Experimental): Patients receive Tarceva 150 mg daily for 21 consecutive days (one treatment cycle). In addition, all patients will receive single agent Taxotere 60 mg/m2 IV over 1 hour infusion every 21 ± 2 days and have it administered on day 1.
  Taxotere + Tarceva to be taken for three cycles past maximal response or until one of the following occurs: 1) a drug-related toxicity requiring discontinuation, 2) disease progression, or 3) for a maximum of 9 cycles.
  Upon completion of 9 cycles of Taxotere plus Tarceva, patients showing evidence of objective response (CR, PR or stable disease) may continue in the extension phase of the study and receive treatment with Tarceva alone. Treatment response evaluated after four cycles of Tarceva treatment(immediately prior to cycle 14). Patients with progression of disease will be taken off study. Responding and stable disease patients will remain on study for up to 8 extension-phase cycles for a total of 17 cycles.
  Interventions: Drug: docetaxel; Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: docetaxel — Administered as an IV infusion of 60m/m2 over a 1-hour period, once every 21 ± 2 days
  Other Names: Taxotere
Drug: erlotinib hydrochloride — Will be taken at a starting daily dose of 150mg
  Other Names: Tarceva

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining docetaxel with erlotinib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with erlotinib works in treating older patients with progressive prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate and response duration in older patients with progressive hormone refractory prostate cancer treated with docetaxel and erlotinib.

Secondary

* Determine the safety of this regimen in these patients.
* Evaluate the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Initial combination therapy: Patients receive docetaxel IV over 1 hour on day 1 and oral erlotinib once daily on days 1-21. Treatment repeats every 21 days for up to 9 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease receive 3 additional courses beyond maximal response.
* Extension phase: After 9 courses of initial combination therapy, patients achieving a complete response, partial response, or stable disease receive 8 courses of erlotinib alone (total of 17 courses of study treatment).

Quality of life is assessed at baseline, day 1 of each course, and at the end of study treatment. For patients in the extension phase, quality of life is also assessed on day 1 of courses 10, 12, 14, and 16.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 22 patients will be accrued for this study within 24 months.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed adenocarcinoma of the prostate.
* Disease progression following primary or secondary hormonal therapy.
* All patients must be maintained on GnRH analog during this study.
* Serum PSA must be > 20 ng/mL in patients without bidimensionally measurable disease or bone disease.
* Age > 65 years.
* Karnofsky performance status of > 70%.
* Life Expectancy of > 12 weeks.
* Peripheral neuropathy, if present must be < grade 1 by NCI criteria.
* Radionuclide bone scan and chest /abdominal/pelvic CT scan must be obtained in all patients within 4 weeks prior to cycle 1/day 1.
* Sexually active men must be willing to consent to using effective contraception while on treatment and for 6 months following treatment.
* No concomitant use of prostata or saw palmetto.
* Testosterone must be castrate levels(< 50 ng/ml).
* WBC > 2.8 x 109/L
* Granulocytes > 1.5 x 109/L
* Platelets > 100 x 109/L
* Hemoglobin > 8.0 g/dL
* Serum creatinine < 2.1
* Total bilirubin < ULN
* Alkaline Phosphatase < 2.5 ULN AND ALT/AST < 2.0 ULN OR Alkaline Phosphatase 2.6-3.9 ULN, AND ALT/AST <1.5 ULN OR Patients with known bone involvement may be included with alkaline phosphatase > 4.0 ULN, IF ALT and AST and total bilirubin are within the normal range and the bone involvement is thought to account for elevated alkaline phosphatase.
* PT, INR should be within physiologic limits, i.e. INR 0.7 - 1.5. If patient is receiving anticoagulation therapy then INR should be within the range of 2.0 - 3.5.

Exclusion Criteria

* Any major surgery or radiotherapy, within 4 weeks prior to cycle 1/day 1 (within 12 weeks for previous treatment with strontium-89, rhenium, or sumarium).
* Hormonal therapy, with the exception of androgen deprivation therapy and stable regimens of prednisone and dexamethasone, (no change within 2 weeks prior to cycle1/day 1). Prior prostate hormonal treatment must have been discontinued at least four weeks (6 weeks for Casodex) prior to cycle1/day 1.
* Cardiovascular: Uncontrolled hypertension (resting blood pressure >160/100 mm/Hg); clinical episodes of congestive heart failure, angina pectoris, or myocardial infarction within the last year.
* Any active infections (requiring IV antibiotics).
* Any prior chemotherapy.
* Not reliable for adequate follow-up.
* History of severe hypersensitivity reaction to drugs formulated with polysorbate 80.
* Brain metastases or (clinical signs of) brain involvement or leptomeningeal disease.
* Patients with a history of another malignancy during the last 5 years other than prostate cancer, nonmelanomatous skin cancer or in situ bladder cancer (Stage T1a).
* Concurrent commercial or investigational antineoplastic therapy.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2004-05; Primary Completion 2006-06 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Response | 9 weeks
  During the primary phase of the study (cycles 1-9), response to the combination of Taxotere® and Tarceva™ treatment will be assessed at the end of every 3 treatment cycles (9 weeks) with the standard procedures such as physical examination, CT scans, bone scans, MRI and laboratory results. For those patients that continue on in the extension phase of the study (cycles 10 -17), response to Tarceva™ is to be assessed at the end of 4 treatment cycles (end of cycle 13).

SECONDARY OUTCOMES:
Safety and tolerability based on adverse events, laboratory tests and physical exams | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allan Pantuck, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington